CLINICAL TRIAL: NCT04107077
Title: A Phase IIa Study of Laparoscopic Hyperthermic Intraperitoneal Chemotherapy (HIPEC) and PD-L1 Expression in Gastric Cancer With Peritoneal Metastases
Brief Title: Phase II Study of the Effects of Laparoscopic Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Patients With Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-0160
Record Dates: First submitted 2019-09-18; First posted 2019-09-27 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer; Peritoneal Carcinomatosis
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms | interventions — Cisplatin; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug Administration Period (Experimental)
  Interventions: Drug: Cisplatin; Drug: Mitomycin

INTERVENTIONS:
Drug: Cisplatin — Laparoscopic HIPEC will be performed at a maximum of two (2) times spaced approximately 6 weeks apart. The dosing of the drugs will be the same during each administration but adjusted if needed based on lab work. The typical dosages are 200mg of Cisplatin
Drug: Mitomycin — Laparoscopic HIPEC will be performed at a maximum of two (2) times spaced approximately 6 weeks apart. The dosing of the drugs will be the same during each administration but adjusted if needed based on lab work. The typical dosages are 30mg of Mitomycin C.

SUMMARY:
To assess if PD-L1 expression can be upregulated in peritoneal metastases from gastric cancer after the administration of HIPEC with greater frequency compared to systemic chemotherapy alone

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed GC/PM only and/or positive peritoneal cytology, who have completed prior systemic chemotherapy for a minimum of 2 to 4 months duration.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of HIPEC for GC/PM in patients under 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Patients must have adequate organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
  * creatinine ≤ institutional ULN OR
  * glomerular filtration rate (GFR) ≥50 mL/min/1.73 m2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m2 (see Appendix B).
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Expected survival greater than 3 months.
* Because cisplatin and Mitomycin C are pregnancy category D and potentially teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of the study.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with coexistence of another untreated malignant neoplasm other than basal cell carcinoma of the skin within the last five years.
* Sites of metastases other than loco-regional lymph nodes and peritoneum (ex. Visceral metastases such as liver, lungs, bone, brain).
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Patients who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin and Mitomycin C.
* Patients with uncontrolled intercurrent illness.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because cisplatin and Mitomycin C are class D agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cisplatin and Mitomycin C, breastfeeding should be discontinued if the mother is treated with cisplatin and Mitomycin C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The PD-L1 expression can be upregulated after administration of HIPEC with greater frequency | 2 years
  To examine if PD-L1 expression can be upregulated in peritoneal metastases from gastric cancer after the administration of HIPEC with greater frequency compared to systemic chemotherapy alone. PD-L1 expression will be measured quantitatively by combined positive score (CPS), with upregulation defined as an quantitative increase in PD-L1 expression via CPS compared to the previously measured timepoint (baseline CPS of 0).

SECONDARY OUTCOMES:
The rate of conversion to resectability with repeated interval laparoscopic HIPEC | 2 years
  To examine the rate of conversion to resectability with repeated interval laparoscopic HIPEC as defined by the Phase II trial published by Badgwell et al.
To quantitatively assess peritoneal cancer index (PCI) change with repeated interval laparoscopic HIPEC. | 2 years
  To quantitatively assess peritoneal cancer index (PCI) change with repeated interval laparoscopic HIPEC.
Overall Survival Rate | 2 years
  To examine overall survival from diagnosis of metastatic disease. Given the potential for longer survival with repeated interval laparoscopic HIPEC compared to systemic chemotherapy alone, this metric will be assessed. In addition, in (+)PD-L1 patients, survival data in this population undergoing repeated interval laparoscopic HIPEC and systemic PD-1 inhibition is unknown.
Perioperative morbidity at 30 days | 30 days
  To assess perioperative morbidity at 30 days.
Perioperative mortality at 30 days | 30 days
  To assess perioperative mortality at 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ardaman Shergill, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States